CLINICAL TRIAL: NCT00272259
Title: Robots for Stroke Survivors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: NSF 0238204
Record Dates: First submitted 2006-01-03; First posted 2006-01-05 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Procedure: Participants will interact with up to two small robots and a visual display

SUMMARY:
The investigators are looking for individuals who have suffered a stroke to participate in an experiment examining the use of robotics in rehabilitation. They are trying to develop a robotic environment for hands after having had a stroke. Participants will interact with up to two small robots and a visual display. The experiment involves minimal risk and may involve testing sessions over multiple weeks. Subjects must be at least 1 year post-stroke and have difficulty picking up small objects.

For more information, contact: Bambi Brewer, CMU Ph.D. Student, 412-241-9423 or bambi@andrew.cmu.edu.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 year post-stroke
* Difficulty picking up small objects

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yoky Matsuoka, Ph.D., Principal Investigator — Carnegie Mellon University; Roberta Klatzky, Ph.D., Study Director — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States